CLINICAL TRIAL: NCT00577733
Title: Pathophysiological Study of Obesity-related Asthma
Brief Title: Study of the Physiology of the Asthma of the Obese Subjects. Breathing Obesity Asthma Study (BOA)
Acronym: BOA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P061010
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2007-12

CONDITIONS: Asthma; Obesity
Keywords: Pulmonary function test; Methacholine challenge; Breathing variability; Polygraphy
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- obese: obese
- healthy volunteers: healthy volunteers

SUMMARY:
Asthma is more frequent in obese women, but the mechanisms underlying the causes of this increased frequency are unknown and are different from usual asthma pathophysiology (associated with allergy). Obesity is known to influence ventilation; our hypothesis is that the normal variability of ventilation is decreased in obese patients, and that this decrease is responsible for an increased reactivity of their airway to non specific stimuli. In this observational study, breathing variability will be studied using polygraphy (an investigation that is made in these women to detect nocturnal apneas), and airway reactivity is studied between pulmonary function tests that are made before bariatric surgery.

DETAILED DESCRIPTION:
Background : An increase in asthma prevalence (or asthma-like symptoms) has been established in obese subjects, especially women. The aim of this pathophysiological study is to evaluate whether the modifications of respiratory mechanics due to severe obesity (Body Mass Index [BMI]>35) may explain the increase in asthma prevalence. Our hypothesis is that a decrease in variability of tidal breathing (evaluated by the coefficient of variation of Tidal volume: CVTV) (which traduces a physiological response to the increased work of breathing) associated with a decrease in the frequency of deep inhalations (FDI) (physiological sighs). The bronchodilatory and bronchoprotective roles of these deep inhalations have been demonstrated. The avoidance of deep inhalations during 10 minutes in healthy subjects is responsible for a non specific transient airway hyperresponsiveness (AHR) to methacholine. Consequently, obesity-related asthma could be due to the loss of bronchoprotective effect of deep inhalations.

Aims: The aim of this study is to evaluate whether 1) the variability of their diurnal ventilation (based on the measurement of CVTV and FDI) in three groups of women: obese with AHR, obese without AHR and healthy non obese (main objective), 2) obesity-related asthma pathophysiology is linked to atopy, and 3) obese asthmatic women have a greater decrease in ventilation variability as compared to non asthmatic obese women (secondary objectives).

Methods: The prevalence of AHR and confirmed asthma (international clinical and functional definition) are determined based on pulmonary function test (spirometry, volume determinations, arterial blood gas, measurement of the resistance of the respiratory system with evaluation of the response to deep inhalation, methacholine challenge, exhaled NO measurement, nocturnal polygraphy and oeso-gastroscopy) results obtained from 150 obese (BMI > 35). The FDI and CVTV will be determined based on the tidal volume obtained from thoracic and abdominal plethysmography inductance measurements during the polygraphy. A nocturnal polygraphy is systematically done in these women to search for a Sleep Apnea Syndrome. 30 healthy (non asthmatic, normal exhaled NO value, BMI 18.5 to 25) women will constitute a control group. The size of the groups have been calculated based on literature data concerning the FDI and CVTV.

Analysis criteria: The prevalences of asthma (or asthma-like symptoms) and AHR will be of 30% and 50% (based on a personal preliminary study), respectively. The FDI and CVTV will be compared in obese women with and without AHR and in healthy women (primary objective), and subsequently in obese asthmatic women and obese non asthmatic women. The measurement of exhaled NO and the bronchomotor effect of deep inhalation will allow the determination of underlying pathophysiology of obesity-related asthma (secondary objective).

Perspectives: If our hypothesis is verified, obesity treatment will become part of the management of asthma in women.

ELIGIBILITY:
Inclusion Criteria:

* female
* age>18 and < 55 years
* BMI>35 (< 25 for healthy women)
* planned bariatric surgery

Exclusion Criteria:

* sleep apnea syndrome
* pregnant or breast-feeding women
* No affiliation or non beneficiary of the National Health Insurance

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: obese with AHR, obese without AHR and healthy non obese
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
compare the variability of the diurnal ventilation (based on the measurement of CVTV and FDI) in three groups of women: obese with AHR, obese without AHR and healthy non obese. | 24 hours

SECONDARY OUTCOMES:
evaluate if the obesity-related asthma pathophysiology is linked to atopy, and if obese asthmatic women have a greater decrease in ventilation variability as compared to non asthmatic obese women | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: DELCLAUX MD Christophe, PhD, Principal Investigator — Department of Physiology, Hôpital Européen Georges Pompidou
Locations (1):
- Department of Physiology, Hôpital Européen Georges Pompidou, Paris, France